CLINICAL TRIAL: NCT00906672
Title: Medico Economic Evaluation of Dermal Substitute Integra® for Coverage of Inferior Limb Traumatic Skin Loss
Acronym: INTEGRA®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2008/26
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Leg Injuries; Ankle Injuries; Foot Injuries
Keywords: Dermal substitute Integra®; Flap; graft; traumatic wound; medico economic costs; esthetical and functional scar results
MeSH Terms: conditions — Leg Injuries; Ankle Injuries; Foot Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- INTEGRA® (Experimental)
  Interventions: Device: INTEGRA®
- Flap technique (Active Comparator)
  Interventions: Procedure: Flap technique

INTERVENTIONS:
Device: INTEGRA® — A plaque of dermal substitute Integra® is adjusted to the size of the wound and sutured. A negative pressure bandage is placed on the wound. 7 to 11 days post surgery, the Integra® silicone layer is removed and the neoderm is covered with a skin graft.
  Arms: INTEGRA®
Procedure: Flap technique — A flap is a part of skin, cutaneous tissue or muscle that is taken from an healthy area of the body and put on the damaged area for coverage.
  Arms: Flap technique

SUMMARY:
Comparison of 2 techniques of surgery on patients with inferior limb traumatic wounds: the innovative technique Integra® and the technique of reference: the flap surgery.

DETAILED DESCRIPTION:
Traumatic skin loss with bone or tendon exposure essentially affects inferior limbs. There are considered serious as they often lead to functional and esthetical consequences, and they generally affect young people.

Flap surgery is the treatment of reference for these skin losses. This technique requires expensive material and a lot of medical staff. The intervention and duration of hospitalisation are often long with heavy medication. Post surgery complications or disabling sequelea involve surgical re-interventions which increase duration of hospital stay and medical staff availability.

The dermal substitute Integra® (Integra LifeSciences Corporation) is an advanced wound care device comprised of a porous matrix of cross-linked bovine tendon collagen and glycosaminoglycan and a semi-permeable polysiloxane (silicone layer). This medical device allows formation of a neoderm. The silicon layer is a temporary layer which is removed when the neoderm is totally built. This surgery is fast, non-invasive, with short hospital stay and limited complications which can be treated easily.

Objective of the study: to assess medico-economic interest of innovative surgery using dermal substitute Integra® compared to the reference using flap surgery in the treatment of traumatic skin loss of inferior limbs. Assessment will be based on re-interventions incidence, long-term functional and esthetical scar results and total cost of each technique.

Study design: multicenter, randomized, open label, parallel design, clinical trial in 12 French plastic surgery / burn care centres.

Planned number of enrolled patients: 120 (80 patients receiving Integra® and 40 patients receiving the flap surgery). Patients will be randomized in 1 of the 2 groups, with an imbalance in favour of the innovative technique.

Duration of enrollment: 24 months Duration of patient follow up: 18 months

ELIGIBILITY:
Inclusion Criteria:

* patient with skin loss traumatic or chronic wound
* wound located from mid third of the leg to distal extremity of feet
* with muscle and/or tendon and/or bone and/or articulation exposure
* requiring a first surgical intervention for the coverage of the skin loss
* patient eligible to the Integra® surgery techniques
* patient with social security affiliation
* written informed consent signed by the patient or representative

Exclusion Criteria:

* Bone fracture located in the skin loss
* Non traumatic wound
* Wound with muscle exposure only
* Immunocompromised patient
* Allergy to bovine collagen, glycosaminoglycans or silicon
* patient with an healthstate that compromise the 18 months Follow-up
* pregnant women / who intend to become pregnant within the 18 months of follow-up
* Patient under administrative or legal supervision

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of at least one complication requiring a surgical re-intervention | Within the first 18 months after surgery
Persistence of an important / major trouble of the scar measured by a "scar-trouble scale" filled in by the patient. | at 18 month-follow up
Auto-evaluation of patient's scar esthetical result with a visual analog scale. | at 18 month-follow up

SECONDARY OUTCOMES:
Occurrence of all post surgical complications | Within the first 18 months after surgery
Duration of hospitalization and healing | Within the first 18 months after surgery
Period until return to work and re-start of daily activities | Within the first 18 months after surgery
Ïntensity of scar pain during cares evaluated with a visual analog scale and quality of life (EuroQol) | Within the first 18 months after surgery
Human and medical requirements | Within the first 18 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Geneviève CHENE, MD-PHD, Study Chair — USMR (University Hospital, Bordeaux); Vincent CASOLI, MD-MHD, Study Director — University Hospital, Bordeaux
Locations (7):
- France (7):
  - University Hospital, Besançon
  - Universiy Hospital Bordeaux,, Bordeaux
  - University Hospital, Clermont-Ferrand
  - University Hospital, Grenoble
  - University Hospital, Montpellier
  - Saint Roch Hospital, Nice
  - University Hospital, Pointe à Pitre